CLINICAL TRIAL: NCT00195715
Title: A Multi Center, Open Label Study of the Human Anti TNF Monoclonal Antibody Adalimumab to Evaluate the Long Term Safety and Tolerability of Repeated Administration of Adalimumab in Subjects With Crohn's Disease
Brief Title: Long-term Safety and Tolerability Study of Adalimumab in Subjects With Crohn's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Mary Beth Tighe Associate Director, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M04-690
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2010-01-07 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Adalimumab 40 mg by subcutaneous injection every other week or every week
  Other Names: ABT-D2E7; Humira

SUMMARY:
To evaluate the long-term maintenance of response, safety and tolerability of repeated administration of adalimumab in subjects with Crohn's disease who participated in and successfully completed Protocol M02-404 or Protocol M04-691.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have successfully completed either the M02-404 (NCT00077779) or M04-691 (NCT00105300) protocol to be eligible for this study
* Diagnosis of Crohn's disease
* Willing and able to give informed consent

Exclusion Criteria:

* Diagnosis of ulcerative colitis
* Women cannot be pregnant or breastfeeding
* Previous history of listeria infection or untreated tuberculosis
* Previous history of cancer other than successfully treated skin cancer or carcinoma-in-situ of the cervix

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 777 (Actual)
Dates: Start 2004-09; Primary Completion 2006-03 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Camez, MD, Study Director — Abbott
Locations (111):
- United States (63):
  - Site Ref # / Investigator 1894, Huntsville, Alabama
  - Site Ref # / Investigator 1895, Jacksonville, Alabama
  - Site Ref # / Investigator 1787, La Jolla, California
  - Site Ref # / Investigator 1902, Roseville, California
  - Site Ref # / Investigator 1824, San Diego, California
  - Site Ref # / Investigator 1891, San Diego, California
  - Site Ref # / Investigator 1860, Englewood, Colorado
  - Site Ref # / Investigator 6178, Lone Tree, Colorado
  - Site Ref # / Investigator 1904, Wheat Ridge, Colorado
  - Site Ref # / Investigator 1858, Bridgeport, Connecticut
  - Site Ref # / Investigator 1827, Clearwater, Florida
  - Site Ref # / Investigator 1883, Gainesville, Florida
  - Site Ref # / Investigator 1909, Hollywood, Florida
  - Site Ref # / Investigator 1884, Ormond Beach, Florida
  - Site Ref # / Investigator 1786, Winter Park, Florida
  - Site Ref # / Investigator 1912, Atlanta, Georgia
  - Site Ref # / Investigator 1878, Arlington Heights, Illinois
  - Site Ref # / Investigator 2534, Chicago, Illinois
  - Site Ref # / Investigator 1823, Peoria, Illinois
  - Site Ref # / Investigator 1885, Anderson, Indiana
  - Site Ref # / Investigator 1900, Indianapolis, Indiana
  - Site Ref # / Investigator 1890, Indianapolis, Indiana
  - Site Ref # / Investigator 1892, Lexington, Kentucky
  - Site Ref # / Investigator 1906, Metairie, Louisiana
  - Site Ref # / Investigator 1881, Annapolis, Maryland
  - Site Ref # / Investigator 1829, Chevy Chase, Maryland
  - Site Ref # / Investigator 1782, Lutherville, Maryland
  - Site Ref # / Investigator 1887, Silver Spring, Maryland
  - Site Ref # / Investigator 2602, Worcester, Massachusetts
  - Site Ref # / Investigator 1773, Plymouth, Minnesota
  - Site Ref # / Investigator 1856, Rochester, Minnesota
  - Site Ref # / Investigator 1832, Jackson, Mississippi
  - Site Ref # / Investigator 1880, Kansas City, Missouri
  - Site Ref # / Investigator 1853, Mexico, Missouri
  - Site Ref # / Investigator 1888, St Louis, Missouri
  - Site Ref # / Investigator 1862, St Louis, Missouri
  - Site Ref # / Investigator 1901, Egg Harbor, New Jersey
  - Site Ref # / Investigator 1825, Great Neck, New York
  - Site Ref # / Investigator 1848, Lake Success, New York
  - Site Ref # / Investigator 1841, New York, New York
  - Site Ref # / Investigator 1852, Asheville, North Carolina
  - Site Ref # / Investigator 1882, Charlote, North Carolina
  - Site Ref # / Investigator 1855, Charlotte, North Carolina
  - Site Ref # / Investigator 1911, Raleigh, North Carolina
  - Site Ref # / Investigator 1861, Wilmington, North Carolina
  - Site Ref # / Investigator 1784, Beachwood, Ohio
  - Site Ref # / Investigator 1896, Beavercreek, Ohio
  - Site Ref # / Investigator 1833, Cincinnati, Ohio
  - Site Ref # / Investigator 1826, Cleveland, Ohio
  - Site Ref # / Investigator 1822, Portland, Oregon
  - Site Ref # / Investigator 1886, Pittsburgh, Pennsylvania
  - Site Ref # / Investigator 1905, Columbia, South Carolina
  - Site Ref # / Investigator 1769, Germantown, Tennessee
  - Site Ref # / Investigator 1907, Nashville, Tennessee
  - Site Ref # / Investigator 1963, Nashville, Tennessee
  - Site Ref # / Investigator 1899, Round Rock, Texas
  - Site Ref # / Investigator 1903, Salt Lake City, Utah
  - Site Ref # / Investigator 6180, Charlottesville, Virginia
  - Site Ref # / Investigator 1783, Danville, Virginia
  - Site Ref # / Investigator 1897, Norfolk, Virginia
  - Site Ref # / Investigator 1850, Spokane, Washington
  - Site Ref # / Investigator 1831, Milwaukee, Wisconsin
  - Site Ref # / Investigator 1849, West Bend, Wisconsin
- Australia (4):
  - Site Ref # / Investigator 1938, Camperdown, New South Wales
  - Site Ref # / Investigator 1940, Bedford Park, South Australia
  - Site Ref # / Investigator 1935, Box Hill, Victoria
  - Site Ref # / Investigator 1937, Parkville, Victoria
- Belgium (3):
  - Site Ref # / Investigator 1941, Bonheiden
  - Site Ref # / Investigator 5189, Brussels
  - Site Ref # / Investigator 2535, Leuven
- Canada (15):
  - Site Ref # / Investigator 1868, Calgary, Alberta
  - Site Ref # / Investigator 1924, Edmonton, Alberta
  - Site Ref # / Investigator 426, Edmonton, Alberta
  - Site Ref # / Investigator 1914, Vancouver, British Columbia
  - Site Ref # / Investigator 1872, Vancouver, British Columbia
  - Site Ref # / Investigator 1870, Victoria, British Columbia
  - Site Ref # / Investigator 1874, Winnipeg, Manitoba
  - Site Ref # / Investigator 1873, Halifax, Nova Scotia
  - Site Ref # / Investigator 1876, Hamilton, Ontario
  - Site Ref # / Investigator 1875, London, Ontario
  - Site Ref # / Investigator 1772, Toronto, Ontario
  - Site Ref # / Investigator 1865, Toronto, Ontario
  - Site Ref # / Investigator 2459, Montreal, Quebec
  - Site Ref # / Investigator 1866, Montreal, Quebec
  - Site Ref # / Investigator 1863, Québec, Quebec
- Denmark (2):
  - Site Ref # / Investigator 1952, Arhus C
  - Site Ref # / Investigator 1922, Odense C
- France (3):
  - Site Ref # / Investigator 1964, Amiens
  - Site Ref # / Investigator 2458, Lillie Cedex
  - Site Ref # / Investigator 1913, Paris
- Germany (3):
  - Site Ref # / Investigator 1942, Kiel
  - Site Ref # / Investigator 2524, Regensburg
  - Site Ref # / Investigator 1943, Stuttgart
- Hungary (2):
  - Site Ref # / Investigator 1944, Budapest
  - Site Ref # / Investigator 1916, Szekszárd
- Italy (3):
  - Site Ref # / Investigator 342, Bologna
  - Site Ref # / Investigator 1945, Rome
  - Site Ref # / Investigator 1779, Turin
- Netherlands (2):
  - Site Ref # / Investigator 1919, Amsterdam
  - Site Ref # / Investigator 1946, Heerlen
- Poland (2):
  - Site Ref # / Investigator 1948, Szczecin, 71-252
  - Site Ref # / Investigator 1947, Warsaw
- South Africa (3):
  - Site Ref # / Investigator 1844, Johannesburg, GT
  - Site Ref # / Investigator 1846, Durban, NL
  - Site Ref # / Investigator 1763, Cape Town, WC
- Spain (2):
  - Site Ref # / Investigator 341, Madrid
  - Site Ref # / Investigator 2457, Port de Sagunt
- Sweden (2):
  - Site Ref # / Investigator 1949, Gothenburg
  - Site Ref # / Investigator 1778, Stockholm
- United Kingdom (2):
  - Site Ref # / Investigator 1951, Edinburgh
  - Site Ref # / Investigator 1771, Rotherham

REFERENCES:
- [Derived] Ryan C, Sobell JM, Leonardi CL, Lynde CW, Karunaratne M, Valdecantos WC, Hendrickson BA. Safety of Adalimumab Dosed Every Week and Every Other Week: Focus on Patients with Hidradenitis Suppurativa or Psoriasis. Am J Clin Dermatol. 2018 Jun;19(3):437-447. doi: 10.1007/s40257-017-0341-6. PMID 29380251
- [Derived] Schreiber S, Reinisch W, Colombel JF, Sandborn WJ, Hommes DW, Robinson AM, Huang B, Lomax KG, Pollack PF. Subgroup analysis of the placebo-controlled CHARM trial: increased remission rates through 3 years for adalimumab-treated patients with early Crohn's disease. J Crohns Colitis. 2013 Apr;7(3):213-21. doi: 10.1016/j.crohns.2012.05.015. Epub 2012 Jun 16. PMID 22704916
- [Derived] Colombel JF, Schwartz DA, Sandborn WJ, Kamm MA, D'Haens G, Rutgeerts P, Enns R, Panaccione R, Schreiber S, Li J, Kent JD, Lomax KG, Pollack PF. Adalimumab for the treatment of fistulas in patients with Crohn's disease. Gut. 2009 Jul;58(7):940-8. doi: 10.1136/gut.2008.159251. Epub 2009 Feb 6. PMID 19201775

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label Adalimumab: 40 mg by subcutaneous injection every other week or every week
Period: Overall Study
Arm/Group | Open-label Adalimumab
Started | 777
Completed | 400
Not Completed | 377
Not completed — Adverse Event | 122
Not completed — Withdrawal by Subject | 58
Not completed — Lost to Follow-up | 27
Not completed — Protocol Violation | 13
Not completed — Lack of Efficacy | 93
Not completed — Pregnancy | 14
Not completed — Investigative site closure | 8
Not completed — Subject moved/relocated | 7
Not completed — Subject non-compliance | 6
Not completed — Subject started commercial Humira | 5
Not completed — Subject choice | 3
Not completed — Loss of response/no improvement | 3
Not completed — Sponsor stopped study | 1
Not completed — Administrative reasons | 2
Not completed — Investigator's decision | 2
Not completed — Subject wants to get pregnant | 4
Not completed — Use of prohibited medication | 2
Not completed — Planned surgery | 2
Not completed — Increased infection rate | 1
Not completed — Ineligible | 1
Not completed — Colonic stricture | 1
Not completed — Sponsor discontinued trial | 1
Not completed — Sponsor discretion - trial ended early | 1

BASELINE CHARACTERISTICS:
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Age Continuous [Mean (Standard Deviation); unit: years] | 38.0 (11.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 485
  Male | 292
Region of Enrollment [Number; unit: participants]
  United States | 349
  Australia | 40
  Belgium | 66
  Canada | 197
  Denmark | 18
  France | 24
  Germany | 5
  Hungary | 8
  Italy | 9
  Netherlands | 10
  Poland | 12
  South Africa | 20
  Spain | 3
  Sweden | 5
  United Kingdom | 11

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Subjects Achieving Clinical Remission
Description: Clinical remission was defined as a Crohn's Disease Activity Index (CDAI) score of < 150. The CDAI is a weighted composite score of 8 clinical factors measured over a 1-week period. A lower CDAI score indicates lesser disease severity.
Time Frame: Week 48
Population: Intent-to-treat, Observed Cases
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 609
Percentage of participants | 59.4

2. Secondary Outcome: Percentage of Subjects Achieving Clinical Remission
Description: as for outcome 1
Time Frame: Week 108
Population: Intent-to-treat, Observed Cases
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 462
Percentage of participants | 68.8

3. Primary Outcome: Percentage of Subjects Achieving Clinical Remission
Description: as for outcome 1
Time Frame: Week 156
Population: Intent-to-treat, defined as all subjects who received at least 1 dose of study drug; Observed Cases
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 272
Percentage of participants | 69.5

4. Secondary Outcome: Percentage of Subjects Achieving Clinical Remission
Description: as for outcome 1
Time Frame: Week 204
Population: Intent-to-treat, Observed Cases
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 15
Percentage of participants | 46.7

5. Secondary Outcome: Percentage of Subjects Achieving Clinical Response 100 (CR-100)
Description: A CR-100 is a decrease from baseline in CDAI score of 100 or more points. The CDAI is a weighted composite score of 8 clinical factors measured over a 1-week period. A lower CDAI score indicates lesser disease severity.
Time Frame: Week 156
Population: Intent-to-treat, Observed Cases
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 272
Percentage of participants | 85.7

6. Secondary Outcome: Percentage of Subjects Achieving Clinical Response 70 (CR-70)
Description: A CR-70 is a decrease from baseline in CDAI score of 70 or more points. The CDAI is a weighted composite score of 8 clinical factors measured over a 1-week period. A lower CDAI score indicates lesser disease severity.
Time Frame: Week 156
Population: Intent-to-treat, Observed Cases
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 272
Percentage of participants | 91.2

7. Secondary Outcome: Percentage of Subjects Achieving Steroid-free Clinical Remission
Description: Steroid-free remission was achieved if the subject stopped taking steroids before the visit and had a Crohn's Disease Activity Index (CDAI) score of <150. The CDAI is a weighted composite score of 8 clinical factors measured over a 1-week period. A lower CDAI score indicates lesser disease severity.
Time Frame: Week 156
Population: Intent-to-treat, Subjects with steroid use at baseline of preceding study, Observed Cases
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 103
Percentage of participants | 63.1

8. Secondary Outcome: Percentage of Subjects Achieving Steroid-free CR-100
Description: Steroid-free CR-100 was achieved if the subject stopped taking steroids before the visit and had a decrease from baseline in CDAI score of 100 or more points at that visit. The CDAI is a weighted composite score of 8 clinical factors measured over a 1-week period. A lower CDAI score indicates lesser disease severity.
Time Frame: Week 156
Population: Intent-to-treat, Subjects with corticosteroid use at baseline of preceding study, Observed Cases
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 103
Percentage of participants | 74.8

9. Secondary Outcome: Percentage of Subjects With Fistula Remission
Description: Fistula remission was defined as the absence of draining fistulas in subjects with fistula present at the preceding study's baseline visit.
Time Frame: Week 156
Population: Intent-to-treat, Subjects with fistulas present at baseline of the preceding study, Observed Cases
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 43
Percentage of participants | 55.8

10. Secondary Outcome: Percentage of Subjects With Infection
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population, defined as all subjects who received at least 1 dose of study drug
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of participants | 80.2

11. Secondary Outcome: Percentage of Subjects With Serious Infection
Description: Serious infections are infectious adverse events that meet at least one criterion for a serious adverse event (e.g., death, life threatening event, hospitalization) including tuberculosis (TB), bacterial sepsis, invasive fungal infections (e.g., histoplasmosis), and infections due to other opportunistic pathogens.
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of participants | 10.6

12. Secondary Outcome: Percentage of Subjects With Malignancy
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of participants | 4.1

13. Secondary Outcome: Percentage of Subjects With Lymphoma
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of participants | 0.1

14. Secondary Outcome: Percentage of Subjects With Nonmelanoma Skin Cancer
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of participants | 1.8

15. Secondary Outcome: Percentage of Subjects With Malignancy (Excluding Nonmelanoma Skin Cancer and Lymphoma)
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of participants | 2.3

16. Secondary Outcome: Percentage of Subjects With Malignancy (Including Lymphoma, Excluding Nonmelanoma Skin Cancer)
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of participants | 2.4

17. Secondary Outcome: Percentage of Subjects With Injection Site Reaction-related Adverse Event
Description: An injection site reaction is any adverse event corresponding to a preferred term beginning with "injection site" excluding injection site arthritis, injection site movement impairment, injection site photosensitivity, injection site joint effusion, injection site joint inflammation, injection site scab, injection site joint pain, or injection site laceration.
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of participants | 22.8

18. Secondary Outcome: Percentage of Subjects With Opportunistic Infection (Excluding Tuberculosis)
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of participants | 4.9

19. Secondary Outcome: Percentage of Subjects With Congestive Heart Failure
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population
Measure: Number; unit: Percentage of subjects
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of subjects | 0

20. Secondary Outcome: Percentage of Subjects With Demyelinating Disease
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of participants | 0.3

21. Secondary Outcome: Percentage of Subjects With Hepatic-related Adverse Event
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of participants | 8.1

22. Secondary Outcome: Percentage of Subjects With Allergic Reaction-related Adverse Event
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of participants | 2.7

23. Secondary Outcome: Percentage of Subjects With Lupus-like Syndrome
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of participants | 0.4

24. Secondary Outcome: Percentage of Subjects With Hematologic-related Adverse Event
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of participants | 1.5

25. Secondary Outcome: Percentage of Subjects With Fatal Adverse Event
Time Frame: Up to 262 weeks of adalimumab treatment
Population: Safety population
Measure: Number; unit: Percentage of participants
Arm/Group | Open-label Adalimumab
Number analyzed (Participants) | 777
Percentage of participants | 0.3

ADVERSE EVENTS:
Time Frame: Up to 262 weeks of adalimumab treatment (includes adalimumab treatment in previous study)
Arm/Group | Open-label Adalimumab
Serious Adverse Events (participants affected / at risk) | 296/777
Other Adverse Events (participants affected / at risk) | 720/777
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Adalimumab (N=777)
Abdominal abscess (Infections and infestations) | 5
Abdominal adhesions (Gastrointestinal disorders) | 2
Abdominal mass (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 11
Abdominal pain upper (Gastrointestinal disorders) | 3
Abdominal rigidity (Gastrointestinal disorders) | 1
Abdominal sepsis (Infections and infestations) | 1
Abortion induced (Surgical and medical procedures) | 3
Abortion of ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 3
Abscess (Infections and infestations) | 3
Abscess intestinal (Infections and infestations) | 2
Abscess limb (Infections and infestations) | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute pulmonary histoplasmosis (Infections and infestations) | 1
Anaemia (Blood and lymphatic system disorders) | 4
Anal abscess (Infections and infestations) | 15
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anal fistula (Gastrointestinal disorders) | 8
Anal stenosis (Gastrointestinal disorders) | 1
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1
Angina unstable (Cardiac disorders) | 1
Anorectal disorder (Gastrointestinal disorders) | 1
Anxiety (Psychiatric disorders) | 1
Appendicitis (Infections and infestations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthritis infective (Infections and infestations) | 1
Ascites (Gastrointestinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2
Axillary vein thrombosis (Vascular disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Basedow's disease (Endocrine disorders) | 1
Bipolar disorder (Psychiatric disorders) | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bladder prolapse (Renal and urinary disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Breast cellulitis (Infections and infestations) | 1
Breast enlargement (Reproductive system and breast disorders) | 1
Breast hyperplasia (Reproductive system and breast disorders) | 1
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1
Bronchitis (Infections and infestations) | 3
Bursitis (Musculoskeletal and connective tissue disorders) | 1
C-reactive protein increased (Investigations) | 1
Calculus ureteric (Renal and urinary disorders) | 2
Campylobacter infection (Infections and infestations) | 1
Carotid artery disease (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 1
Catheter sepsis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Cerebrovascular accident (Nervous system disorders) | 1
Cervical dysplasia (Reproductive system and breast disorders) | 1
Cervicitis (Infections and infestations) | 1
Chest pain (General disorders) | 1
Chills (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 2
Cholelithiasis (Hepatobiliary disorders) | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Clostridial infection (Infections and infestations) | 2
Clostridium difficile colitis (Infections and infestations) | 2
Coccidioidomycosis (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1
Colonic stenosis (Gastrointestinal disorders) | 3
Colpocele (Reproductive system and breast disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Convulsion (Nervous system disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Crohn's disease (Gastrointestinal disorders) | 92
Cystocele (Reproductive system and breast disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 7
Demyelination (Nervous system disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Depression (Psychiatric disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 2
Drug dependence (Psychiatric disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Endometriosis (Reproductive system and breast disorders) | 1
Enteritis (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 2
Escherichia infection (Infections and infestations) | 1
Faecal volume increased (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Feeling cold (General disorders) | 1
Female genital tract fistula (Reproductive system and breast disorders) | 1
Fistula (Musculoskeletal and connective tissue disorders) | 3
Fistula discharge (Musculoskeletal and connective tissue disorders) | 1
Frequent bowel movements (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastroenteritis (Infections and infestations) | 5
Gastroenteritis viral (Infections and infestations) | 3
Gastrointestinal fistula (Gastrointestinal disorders) | 1
Gastrointestinal obstruction (Gastrointestinal disorders) | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Goitre (Endocrine disorders) | 1
Granuloma annulare (Skin and subcutaneous tissue disorders) | 1
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Haemorrhoids (Gastrointestinal disorders) | 2
Head injury (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 2
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hernia (General disorders) | 3
Herpes zoster (Infections and infestations) | 1
Hidradenitis (Skin and subcutaneous tissue disorders) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Hypersensitivity (Immune system disorders) | 1
Hypertension (Vascular disorders) | 1
Hypoaesthesia (Nervous system disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 1
Ileal perforation (Gastrointestinal disorders) | 1
Ileal stenosis (Gastrointestinal disorders) | 4
Ileus (Gastrointestinal disorders) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 2
Insomnia (Psychiatric disorders) | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1
Intestinal fistula (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 10
Intestinal perforation (Gastrointestinal disorders) | 1
Intestinal stenosis (Gastrointestinal disorders) | 2
Iron deficiency (Metabolism and nutrition disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Jejunal perforation (Gastrointestinal disorders) | 1
Joint contracture (Musculoskeletal and connective tissue disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 2
Lobar pneumonia (Infections and infestations) | 3
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Lumbar radiculopathy (Nervous system disorders) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lupus-like syndrome (Musculoskeletal and connective tissue disorders) | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Mammoplasty (Surgical and medical procedures) | 1
Medical device complication (Injury, poisoning and procedural complications) | 1
Medical device removal (Surgical and medical procedures) | 1
Megacolon (Gastrointestinal disorders) | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Menorrhagia (Reproductive system and breast disorders) | 2
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 1
Multiple injuries (Injury, poisoning and procedural complications) | 1
Muscle abscess (Infections and infestations) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Nephrolithiasis (Renal and urinary disorders) | 6
Neuropathy peripheral (Nervous system disorders) | 1
Non-cardiac chest pain (General disorders) | 1
Obstruction (General disorders) | 1
Optic neuritis (Nervous system disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1
Otitis media (Infections and infestations) | 1
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ovarian cyst (Reproductive system and breast disorders) | 5
Overdose (Injury, poisoning and procedural complications) | 1
Pain (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Palpitations (Cardiac disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 2
Pancreatitis acute (Gastrointestinal disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Perineal abscess (Infections and infestations) | 1
Peripheral coldness (General disorders) | 1
Perirectal abscess (Infections and infestations) | 5
Peritonitis (Gastrointestinal disorders) | 1
Peritonsillar abscess (Infections and infestations) | 1
Photophobia (Eye disorders) | 1
Physical assault (Social circumstances) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia (Infections and infestations) | 8
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonia fungal (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 2
Postoperative fever (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 1
Procedural nausea (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Procedural site reaction (Injury, poisoning and procedural complications) | 1
Proctalgia (Gastrointestinal disorders) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary tuberculosis (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 5
Pyrexia (General disorders) | 6
Radius fracture (Injury, poisoning and procedural complications) | 1
Rectal abscess (Infections and infestations) | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1
Rectocele (Reproductive system and breast disorders) | 1
Red blood cell sedimentation rate increased (Investigations) | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal failure acute (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2
Scrotal abscess (Infections and infestations) | 1
Sepsis (Infections and infestations) | 4
Septic shock (Infections and infestations) | 1
Sinus polyp (Respiratory, thoracic and mediastinal disorders) | 1
Sinusitis (Infections and infestations) | 3
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 30
Small intestinal perforation (Gastrointestinal disorders) | 1
Small intestinal stenosis (Gastrointestinal disorders) | 1
Small intestine ulcer (Gastrointestinal disorders) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Staphylococcal infection (Infections and infestations) | 1
Stress urinary incontinence (Renal and urinary disorders) | 1
Substance abuse (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tympanic membrane perforation (Ear and labyrinth disorders) | 1
Urinary tract infection (Infections and infestations) | 3
Urogram normal (Investigations) | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Uterine prolapse (Reproductive system and breast disorders) | 1
Vaginal cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vaginal prolapse (Reproductive system and breast disorders) | 2
Venous thrombosis (Vascular disorders) | 1
Vertebral injury (Injury, poisoning and procedural complications) | 1
Viral infection (Infections and infestations) | 1
Vision blurred (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Vulval abscess (Infections and infestations) | 1
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Weight decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Adalimumab (N=777)
Abdominal distension (Gastrointestinal disorders) | 65
Abdominal pain (Gastrointestinal disorders) | 180
Abdominal pain upper (Gastrointestinal disorders) | 45
Abdominal tenderness (Gastrointestinal disorders) | 45
Anaemia (Blood and lymphatic system disorders) | 46
Anal fistula (Gastrointestinal disorders) | 45
Anxiety (Psychiatric disorders) | 54
Arthralgia (Musculoskeletal and connective tissue disorders) | 192
Back pain (Musculoskeletal and connective tissue disorders) | 87
Bronchitis (Infections and infestations) | 92
Constipation (Gastrointestinal disorders) | 81
Cough (Respiratory, thoracic and mediastinal disorders) | 82
Crohn's disease (Gastrointestinal disorders) | 309
Depression (Psychiatric disorders) | 70
Diarrhoea (Gastrointestinal disorders) | 118
Dizziness (Nervous system disorders) | 54
Dyspepsia (Gastrointestinal disorders) | 64
Eczema (Skin and subcutaneous tissue disorders) | 52
Fatigue (General disorders) | 107
Fistula (Musculoskeletal and connective tissue disorders) | 40
Flatulence (Gastrointestinal disorders) | 44
Gastroenteritis (Infections and infestations) | 58
Gastroenteritis viral (Infections and infestations) | 42
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 54
Headache (Nervous system disorders) | 141
Hypertension (Vascular disorders) | 44
Influenza (Infections and infestations) | 137
Influenza like illness (General disorders) | 48
Injection site irritation (General disorders) | 46
Injection site pain (General disorders) | 43
Injection site reaction (General disorders) | 60
Insomnia (Psychiatric disorders) | 81
Muscle spasms (Musculoskeletal and connective tissue disorders) | 43
Nasopharyngitis (Infections and infestations) | 203
Nausea (Gastrointestinal disorders) | 142
Oedema peripheral (General disorders) | 47
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 84
Pain (General disorders) | 45
Pain in extremity (Musculoskeletal and connective tissue disorders) | 47
Pruritus (Skin and subcutaneous tissue disorders) | 50
Pyrexia (General disorders) | 105
Rash (Skin and subcutaneous tissue disorders) | 100
Sinusitis (Infections and infestations) | 116
Upper respiratory tract infection (Infections and infestations) | 150
Urinary tract infection (Infections and infestations) | 80
Viral infection (Infections and infestations) | 40
Vomiting (Gastrointestinal disorders) | 82

LIMITATIONS AND CAVEATS:
This study was stopped by the sponsor in December 2008 when the pre-specified termination criteria were met. Subjects who continued in the study through the termination date were considered as having completed the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any investigator or institution that plans on presenting/publishing results disclosure, should provide written notification to Abbott within 60 days of their presentation/publication. Abbott requests that no presentation/publication will be allowed until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay of any proposed presentation/publication maybe requested if Abbott needs to secure patent or other proprietary protection.